CLINICAL TRIAL: NCT05799430
Title: Effects of Interdisciplinary Medication Review in Chronic Complex Patients or Patients With Polypharmacy After Hospital Discharge
Brief Title: Medication Review in Chronic Complex or Polymedicated Patients After Hospital Discharge.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Andalusian Health Service (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: S0502
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-04

CONDITIONS: Medication Review; Polypharmacy; Disease, Chronic
Keywords: Medication Review; Polypharmacy
MeSH Terms: conditions — Chronic Disease | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A cluster-randomized control trial
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive a multidisciplinary medication review and a personalized therapeutic plan in the following 72 hours after hospital discharge. The intervention will be developed by a multidisciplinary team that includes a family physician (FP), a primary care nurse (PCN) and a primary care pharmacist (PCP). PCP is a pharmacist working in a full-time base for the Pharmacy Service in a Primary Care District in Andalusian Public Health Service.
  Interventions: Behavioral: Multidisciplinary medication review
- Control group (Active Comparator): The control group will receive usual care.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Multidisciplinary medication review — FP communicate to the PCP patients recently discharged. The medication review process consists in 5 steps:
  1. PCP perform a structured drug review based on information from health record and e-prescribing application. The drug review comprise the appraisal of potentially inappropriate medication based on lists of explicit criteria.
  2. PCP communicates and discuss the results of medication review with GP and PCN, in a brief meeting face-to-face, with possible adaptation of the recommendations.
  3. FP, PCN and PCP agree on a personalized therapeutic plan for the patient that includes actions to optimize the therapy.
  4. FP and PCN share plan with the patient and/or carer with possible adaptation of the recommendations and agree about actions to be implemented.
  5. FP and PCN communicate to PCP final agreement with patient and/or carer
  6. FP and/or PCN follow-up implantation of agreed recommendations using standard health care procedures
  Arms: Intervention
Behavioral: Control group — Usual care by FP an PCN
  Arms: Control group

SUMMARY:
The goal of this prospective multicentre clustered randomized controlled trial is to evaluate the effect on new hospitalization episodes of a multidisciplinary medication review in primary care patients with polypharmacy or chronic complex conditions after hospital discharge.

The multidisciplinary team will be integrated by a family physician (FP), a primary care nurse (PCN) and a primary care pharmacist (PCP). Patient will be adults aged 65 years and older. Polypharmacy refers to the use of 10 or more drugs based on information in electronic prescription software.

Research questions are:

In elderly patients with polypharmacy, which is the effect of an interdisciplinary medication review after hospital discharge in comparison with standard care, in terms of:

* new hospitalization episodes?
* number of drugs prescribed?
* prescribed drugs adequacy?

DETAILED DESCRIPTION:
Centres will be randomized to medication review intervention or usual care group. Eligible patients will be ask for informed consent. For patients in the intervention group, PCP will collect information about prescribed medication and diseases from the electronic health record and e-prescribing application. The medication review in primary care will be focus to reconcile the medications the patient was taking prior to admission and those initiated in hospital, with the medications they should be taking post-discharge to ensure all changes are intentional and that discrepancies are resolved as soon as possible. The review process will include detection of potential drugs interactions, wrong doses, lack of adherence (based on dispensing recorded data) and adequacy to explicit criteria for potentially inappropriate prescriptions included in different tools: a) STOPP-STAR, STOPP-Pal, LESS-CHRON lists; b) Guideline for Medication Review in Primary Care, a local publication and c) Medication review in patients with polypharmacy. A list of drugs frequently associate with potentially inappropriate prescriptions. Andalusian health Service). PCP will write a report to communicate the results of medication review to primary care physician and nurse. The multidisciplinary team will define a personalized therapeutic plan to be implemented for every patient.

Patients in the control group will receive usual care.

ELIGIBILITY:
Inclusion Criteria:

- Hospital discharge in the last 48 h and one of the following conditions:

* Polypharmacy: ten o more drugs prescribed in a chronic schedule OR
* Complez Chronic Condition

Exclusion Criteria:

* Patients in last days of life
* Major mental health disorder
* Patient on dialysis
* Organ transplant patients

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of hospitalization episodes | 12 months
  Registered in Electronic Health Record. In emergency department or in hospital service
Length of Hospital Stay | 12 months
  Registered in Electronic Health Record.

SECONDARY OUTCOMES:
Healthcare utilisation | 12 months
  Number of visits to primary care services (family physician or primary care nurse) and hospital services (non emergency and without hospitalization)
Mortality | 12 month
  Dead for any cause
Number of potentially inappropriate drugs | 12 months
  Total number of potentially inappropriate prescribed drugs based on explicit criteria
Number of medications | 12 months
  Total number of drugs chronically prescribed (treatment length: unless 120 days)
Number of proposal about treatment improvement | 7 days
  Number of proposal about treatment improvement included in PCP report
Number of proposal about treatment improvement agreed with primary care team | 7 days
  Number of proposal about treatment improvement agreed with primary care team in a face face meeting
Number of proposal about treatment improvement accepted by the patient or care | 7 days
  Number of proposal about treatment improvement agreed with primary care team in a face face meeting

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Molina, Pharm Dr, Principal Investigator — Andalusian Health Service. Spain
Locations (1):
- Sevilla Primary Care District, Seville, Spain

REFERENCES:
- [Background] Franchi C, Nobili A, Mari D, Tettamanti M, Djade CD, Pasina L, Salerno F, Corrao S, Marengoni A, Iorio A, Marcucci M, Mannucci PM; REPOSI Investigators. Risk factors for hospital readmission of elderly patients. Eur J Intern Med. 2013 Jan;24(1):45-51. doi: 10.1016/j.ejim.2012.10.005. Epub 2012 Nov 8. PMID 23142413
- [Background] Weinberger M, Oddone EZ, Henderson WG. Does increased access to primary care reduce hospital readmissions? Veterans Affairs Cooperative Study Group on Primary Care and Hospital Readmission. N Engl J Med. 1996 May 30;334(22):1441-7. doi: 10.1056/NEJM199605303342206. PMID 8618584
- [Background] Graham H, Livesley B. Can readmissions to a geriatric medical unit be prevented? Lancet. 1983 Feb 19;1(8321):404-6. doi: 10.1016/s0140-6736(83)91513-1. PMID 6130389
- [Background] Jencks SF, Williams MV, Coleman EA. Rehospitalizations among patients in the Medicare fee-for-service program. N Engl J Med. 2009 Apr 2;360(14):1418-28. doi: 10.1056/NEJMsa0803563. PMID 19339721
- [Background] Acosta-Garcia H, Alfaro-Lara ER, Sanchez-Fidalgo S, Sevilla-Sanchez D, Delgado-Silveira E, Juanes-Borrego A, Santos-Ramos B. Intervention effectiveness by pharmacists integrated within an interdisciplinary health team on chronic complex patients. Eur J Public Health. 2020 Oct 1;30(5):886-899. doi: 10.1093/eurpub/ckz224. PMID 32052027
- [Background] Guisado-Gil AB, Mejias-Trueba M, Alfaro-Lara ER, Sanchez-Hidalgo M, Ramirez-Duque N, Santos-Rubio MD. Impact of medication reconciliation on health outcomes: An overview of systematic reviews. Res Social Adm Pharm. 2020 Aug;16(8):995-1002. doi: 10.1016/j.sapharm.2019.10.011. Epub 2019 Oct 17. PMID 31883776
- [Background] Santos-Ramos B, Otero Lopez MJ, Galvan-Banqueri M, Alfaro-Lara ER, Vega-Coca MD, Nieto-Martin MD, Ollero-Baturone M. [Health care models for patients with multiple chronic conditions and the role of the hospital pharmacy/the hospital pharmacist]. Farm Hosp. 2012 Nov-Dec;36(6):506-17. doi: 10.7399/FH.2012.36.6.52. Spanish. PMID 23461444
- [Background] Alfaro-Lara ER, Vega-Coca MD, Galvan-Banqueri M, Nieto-Martin MD, Perez-Guerrero C, Santos-Ramos B. [Pharmacological treatment conciliation methodology in patients with multiple conditions]. Aten Primaria. 2014 Feb;46(2):89-99. doi: 10.1016/j.aprim.2013.07.002. Epub 2013 Sep 12. Spanish. PMID 24035767
- [Background] Rodriguez-Perez A, Alfaro-Lara ER, Sierra-Torres MI, Villalba-Moreno A, Nieto-Martin MD, Galvan-Banqueri M, Santos-Ramos B. Validation of the LESS-CHRON criteria: reliability study of a tool for deprescribing in patients with multimorbidity. Eur J Hosp Pharm. 2019 Nov;26(6):334-338. doi: 10.1136/ejhpharm-2017-001476. Epub 2018 May 30. PMID 31798857
- [Background] Rankin A, Cadogan CA, Patterson SM, Kerse N, Cardwell CR, Bradley MC, Ryan C, Hughes C. Interventions to improve the appropriate use of polypharmacy for older people. Cochrane Database Syst Rev. 2018 Sep 3;9(9):CD008165. doi: 10.1002/14651858.CD008165.pub4. PMID 30175841
- [Background] Frazier SC. Health outcomes and polypharmacy in elderly individuals: an integrated literature review. J Gerontol Nurs. 2005 Sep;31(9):4-11. doi: 10.3928/0098-9134-20050901-04. PMID 16190007
- [Background] Fulton MM, Allen ER. Polypharmacy in the elderly: a literature review. J Am Acad Nurse Pract. 2005 Apr;17(4):123-32. doi: 10.1111/j.1041-2972.2005.0020.x. PMID 15819637
- [Background] Shrank WH, Polinski JM, Avorn J. Quality indicators for medication use in vulnerable elders. J Am Geriatr Soc. 2007 Oct;55 Suppl 2:S373-82. doi: 10.1111/j.1532-5415.2007.01345.x. No abstract available. PMID 17910560
- [Background] Cardenas Valladolid J, Mena Mateo J, Canada Dorado MM, Rodriguez Morales D, Sanchez Perruca L. [Implementation and improvement in a care program for the elderly on multiple medications in a primary care area]. Rev Calid Asist. 2009 Feb;24(1):24-31. doi: 10.1016/S1134-282X(09)70072-7. Epub 2009 Feb 23. Spanish. PMID 19369139
- [Background] Weber V, White A, McIlvried R. An electronic medical record (EMR)-based intervention to reduce polypharmacy and falls in an ambulatory rural elderly population. J Gen Intern Med. 2008 Apr;23(4):399-404. doi: 10.1007/s11606-007-0482-z. PMID 18373136
- [Background] Lenaghan E, Holland R, Brooks A. Home-based medication review in a high risk elderly population in primary care--the POLYMED randomised controlled trial. Age Ageing. 2007 May;36(3):292-7. doi: 10.1093/ageing/afm036. Epub 2007 Mar 26. PMID 17387123
- [Background] Hanlon JT, Weinberger M, Samsa GP, Schmader KE, Uttech KM, Lewis IK, Cowper PA, Landsman PB, Cohen HJ, Feussner JR. A randomized, controlled trial of a clinical pharmacist intervention to improve inappropriate prescribing in elderly outpatients with polypharmacy. Am J Med. 1996 Apr;100(4):428-37. doi: 10.1016/S0002-9343(97)89519-8. PMID 8610730
- [Background] Denneboom W, Dautzenberg MG, Grol R, De Smet PA. Treatment reviews of older people on polypharmacy in primary care: cluster controlled trial comparing two approaches. Br J Gen Pract. 2007 Sep;57(542):723-31. PMID 17761060
- [Background] Kirwin JL, Cunningham RJ, Sequist TD. Pharmacist recommendations to improve the quality of diabetes care: a randomized controlled trial. J Manag Care Pharm. 2010 Mar;16(2):104-13. doi: 10.18553/jmcp.2010.16.2.104. PMID 20178395
- [Background] Parody Rua E, Segu Tolosa J. [Cost-effectiveness and cost calculation in an intervention on medication-related problems in primary care]. Aten Primaria. 2005 May 31;35(9):472-7. doi: 10.1157/13075471. Spanish. PMID 15919021
- [Background] Molina Lopez T, Dominguez Camacho JC, Palma Morgado D, Caraballo Camacho Mde L, Morales Serna JC, Lopez Rubio S. [A review of the medication in polymedicated elderly with vascular risk: a randomised controlled trial]. Aten Primaria. 2012 Aug;44(8):453-60. doi: 10.1016/j.aprim.2011.09.015. Epub 2012 Feb 16. Spanish. PMID 22341703
- [Background] Wessell AM, Nietert PJ, Jenkins RG, Nemeth LS, Ornstein SM. Inappropriate medication use in the elderly: results from a quality improvement project in 99 primary care practices. Am J Geriatr Pharmacother. 2008 Mar;6(1):21-7. doi: 10.1016/j.amjopharm.2008.02.001. PMID 18396245
- [Background] Denneboom W, Dautzenberg MG, Grol R, De Smet PA. Analysis of polypharmacy in older patients in primary care using a multidisciplinary expert panel. Br J Gen Pract. 2006 Jul;56(528):504-10. PMID 16834876
- [Background] Zermansky AG, Alldred DP, Petty DR, Raynor DK, Freemantle N, Eastaugh J, Bowie P. Clinical medication review by a pharmacist of elderly people living in care homes--randomised controlled trial. Age Ageing. 2006 Nov;35(6):586-91. doi: 10.1093/ageing/afl075. Epub 2006 Aug 12. PMID 16905764
- [Background] Pit SW, Byles JE, Henry DA, Holt L, Hansen V, Bowman DA. A Quality Use of Medicines program for general practitioners and older people: a cluster randomised controlled trial. Med J Aust. 2007 Jul 2;187(1):23-30. doi: 10.5694/j.1326-5377.2007.tb01110.x. PMID 17605699
- [Background] Royal S, Smeaton L, Avery AJ, Hurwitz B, Sheikh A. Interventions in primary care to reduce medication related adverse events and hospital admissions: systematic review and meta-analysis. Qual Saf Health Care. 2006 Feb;15(1):23-31. doi: 10.1136/qshc.2004.012153. PMID 16456206
- [Background] Nieto-Martin MD, De la Higuera-Vila L, Bernabeu-Wittel M, Gonzalez-Benitez MA, Alfaro-Lara ER, Baron-Ramos MA, Montero-Aparicio E, Aparicio-Santos R, Baturone MO; list of researchers involved in the IMPACTO study and their affiliations. A multidisciplinary approach for patients with multiple chronic conditions: IMPACTO study. Med Clin (Barc). 2019 Aug 2;153(3):93-99. doi: 10.1016/j.medcli.2019.01.014. Epub 2019 Mar 8. English, Spanish. PMID 30857796
- [Background] Brehaut JC, Colquhoun HL, Eva KW, Carroll K, Sales A, Michie S, Ivers N, Grimshaw JM. Practice Feedback Interventions: 15 Suggestions for Optimizing Effectiveness. Ann Intern Med. 2016 Mar 15;164(6):435-41. doi: 10.7326/M15-2248. Epub 2016 Feb 23. PMID 26903136
- [Background] Brotons C, Arino D, Borras I, Buitrago F, Gonzalez ML, Kloppe P, Orozco D, Pepio JM, Rodriguez P, Rodriguez AI; Equipo Investigador del Estudio PREseAP. [Evaluation of the efficacy of a comprehensive programme of secondary prevention of cardiovascular disease in primary care: the PREseAP Study]. Aten Primaria. 2006 Mar 31;37(5):295-8. doi: 10.1157/13086317. Spanish. PMID 16595102
- [Background] Cane J, O'Connor D, Michie S. Validation of the theoretical domains framework for use in behaviour change and implementation research. Implement Sci. 2012 Apr 24;7:37. doi: 10.1186/1748-5908-7-37. PMID 22530986
- See also: Estrategia para la seguridad del paciente. Plan estratégico de calidad del Sistema Sanitario Público de Andalucía. Consejería de Salud y Familias. 2019 — https://juntadeandalucia.es/export/drupaljda/EstrategiaISeguridadPaciente_v5.pdf
- See also: Lown Institute. Medication Overload: America's Other Drug Problem. How the drive to prescribe is harming older adults. 2019 — https://lowninstitute.org/wp-content/uploads/2019/08/medication-overload-lown-web.pdf
- See also: Scottish Government Polypharmacy Model of Care Group. Polypharmacy Guidance, Realistic Prescribing. 3ª edition, 2018. Scottish Government — https://www.therapeutics.scot.nhs.uk/wp-content/uploads/2018/09/Polypharmacy-Guidance-2018.pdf
- See also: Medicines Optimization. Quality standard [QS120] NICE. 2016 — https://www.nice.org.uk/guidance/qs120
- See also: Atención a Pacientes Pluripatológicos. Proceso Asistencial Integrado. Consejería de Salud 2018. — https://juntadeandalucia.es/export/drupaljda/salud_5af1956d9925c_atencion_pacientes_pluripatologicos_2018.pdf
- See also: Plan Andaluz de Atención Integrada a Pacientes con Enfermedades Crónicas. Consejería de Salud. 2012 — https://juntadeandalucia.es/export/drupaljda/PlanAtencEECC.pdf